CLINICAL TRIAL: NCT00184535
Title: Muscle Activity "Onset" in the Transversus Abdominis - Simultaneous Recordings by Intramuscular Electromyography and High Frame Rate Ultrasound Imaging.
Brief Title: Recording Methods of Muscle Activity "Onset".
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Other Study IDs: REK 4.2005.885
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Neuromuscular control; Anticipatory motor control; Musculoskeletal Physiologic Processes; Muscle, Skeletal; Ultrasonography; Electromyography
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delayed anticipatory muscle activity response in deep low back and abdominal muscles has been observed in patients with low back pain, indicative of a pathological condition. Muscle activity onset is traditionally recorded by intramuscular electromyography, but there is a need for a less cumbersome recording method in large clinical studies. The purpose of this experimental study is to explore whether high-frame rate m-mode ultrasound and tissue velocity imaging could measure anticipatory muscle responses ("onset") in the abdominal muscles reliably and comparably accurate to intramuscular EMG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 30-65 yrs

Exclusion Criteria:

* recent low back pain
* low back, neck or shoulder pain inflicting work absence or bed rest
* cardiac, rheumatic or other serious illness
* pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women between 30-65 yrs with no recent low back pain
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, PhD, Study Chair — Norw. Univ of Sci and Technol
Locations (1):
- Norwegian University of Science and Technology (NTNU), Nasjonal senter for spinale lidelser, Trondheim, Norway

REFERENCES:
- [Result] Vasseljen O, Dahl HH, Mork PJ, Torp HG. Muscle activity onset in the lumbar multifidus muscle recorded simultaneously by ultrasound imaging and intramuscular electromyography. Clin Biomech (Bristol). 2006 Nov;21(9):905-13. doi: 10.1016/j.clinbiomech.2006.05.003. Epub 2006 Jul 5. PMID 16822599